CLINICAL TRIAL: NCT03260010
Title: Efficacy and Safety of Intravenous Fosfomycin in Prosthetic Joint Infection (PJI) Caused by Staphylococci, Streptococci, Enterococci and Gram-negative Bacilli, Including Mixed Infections and Culture Negative PJI's ("PROOF-Study")
Brief Title: Efficacy and Safety of Intravenous Fosfomycin in Prosthetic Joint Infection
Acronym: PROOF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pro-Implant Foundation (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROOF
Record Dates: First submitted 2017-08-15; First posted 2017-08-24 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2017-08

CONDITIONS: Prosthetic Joint Infection
MeSH Terms: interventions — Fosfomycin

STUDY DESIGN:
Intervention Model Description: In this open prospective interventional clinical study patients with hip, knee or shoulder PJI (as defined below) caused by fosfomycin-susceptible staphylococci, streptococci, enterococci or gram-negative bacilli will be included. After inclusion and PJI-surgery, intravenous fosfomycin will be given 5 g every 8 hours for 1, 2, 3-or -4 weeks according to the pathogen and surgery procedure and generally as a part of the antibiotic combination therapy of the treatment algorithm. This Treatment is followed by oral antibiotics for a total of 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fosfomycin Arm (Experimental): Include intravenous fosfomycin in the treatment of PJI according to predetermined algorithm
  Interventions: Drug: Fosfomycin

INTERVENTIONS:
Drug: Fosfomycin — Infectofos 5 g

SUMMARY:
The PROOF Study is an open prospective interventional non-randomized study which aim is to determine the outcome / effect and safety of fosfomycin in patients with hip, knee or shoulder PJI.

DETAILED DESCRIPTION:
To confirm a non-inferior effect and the safety of the investigated antimicrobial fosfomycin regimen in PJI of the hip, knee or shoulder against an assumed 80% effect (PJI-free proportion within one year for standard antibiotics aside fosfomycin), following a standardized surgical therapy involving retention, one-stage exchange or two-stage exchange (with short or long interval).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been obtained (prior to planned surgical PJI treatment);
2. Subject is ≥18 years of age;
3. Subject has either a culture negative or a culture positive PJI of the hip, knee or shoulder prosthesis: (i) visible purulence of a preoperative aspirate or intraoperative periprosthetic tissue (as determined by the surgeon),or (ii) presence of a sinus tract communicating with the prosthesis, or (iii) acute inflammation in intraoperative permanent tissue sections by histopathology (as determined by the pathologist), or (iv) microbial growth in preoperative joint aspirate, intraoperative periprosthetic tissue or sonication fluid of the removed implant (>50 CFU/ml sonication fluid), or (v) synovial fluid with >2000 leukocytes/μl or >70% granulocytes; or reasonable evidence for a suspected PJI (based on clinical, laboratory, and radiological criteria) to undergo joint surgery to proof the PJI diagnosis (according to standard of care, Zimmerli W et al. NEJM 2004);
4. For culture positive PJI's at least one of the following isolates:

   staphylococci (fosfomycin MHK ≤ 32 mg/ml), streptococci (MHK ≤ 128 mg/ml), enterococci (MHK ≤ 128 mg/ml), fosfomycin susceptible gram-negative bacilli, including also mixed infections with other pathogens (fosfomycin susceptible or not);
5. Subject is planned to/will undergo appropriate surgical procedure following the state of the art PJI treatment algorithm, which includes either debridement & retention of the prosthesis or exchange of the prosthesis. The exchange includes a one-stage exchange, two-stage prosthesis exchange with a short interval (2- 3 weeks) or long interval (6-8 weeks), according to the treatment algorithm;
6. Subject is willing to participate in the study, follow protocol study treatment regimen, and comply with all planned follow-up assessments.

Exclusion Criteria:

1. Allergy or intolerance (or other contraindication) to fosfomycin;
2. Isolation of fungi (molds or yeasts) or mycobacteria;
3. Isolation of one of the following pathogens: staphylococci fosfomycin MHK > 32 mg/ml, streptococci MHK > 128 mg/ml, enterococci MHK > 128 mg/ml , fosfomycin resistant gramnegative bacilli;
4. Severely compromised bone/soft tissue pre or during surgery (if during surgery: exclusion/withdrawal before IMP application);
5. Pregnancy, and/or woman wishing to become pregnant;
6. Breast-feeding;
7. Women of childbearing potential without at least one of the following contraception methods: correctly placed cooper containing or progestin-containing intrauterine device (IUD); female condom used WITH a spermicide (i.e. foam gel, film, cream, or suppository); bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusive procedure (at least till the end of the ambulatory treatment phase);
8. Subject has been previously enrolled in this study or was enrolled in another interventional medicinal product or medical device study in the last 30 days;
9. Subject had prior exposure to fosfomycin within the past 4 weeks;
10. Inability to read and understand the participant's information;
11. Subjects institutionalized by warrant or court order;
12. Employees of the sponsor or an involved CRO;
13. In pre surgery culture negative patients: All isolates unsusceptible to fosfomycin after surgery (exclusion / early withdrawal after surgery);
14. Suspected PJI not proven after surgery (exclusion / early withdrawal after surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Infection cure rate | 1 year
  Proportion of patients free of PJI relapse (i.e. infection cure rate) within 1 year after inclusion. Relapse is defined as new PJI diagnosis more than 4 weeks after the last surgical intervention of the initial 12 week treatment period.

SECONDARY OUTCOMES:
Infection cure rate | 2 years
  Proportion of patients free of Prosthetic Joint-Infection relapse (infection cure rate) within 2 years after inclusion
Proportion of patients with revision | 1 year
  Proportion of patients with revision (surgical intervention with or without prosthesis removal >4 weeks after last surgical intervention of the initial 12 week treatment period)
Proportion of patients with revision due to hematogenous versus non-hematogenous infection | 1 year
  Proportion of patients with revision due to hematogenous (acute onset with duration of symptoms <3 weeks and onset of symptoms is >3 months after last surgery) versus non-hematogenous infection
Proportion of patients with unscheduled early revisions | 1 year
  Proportion of patients with unscheduled early revisions (<4 weeks after last scheduled surgical intervention - deep (= bone/joint) revision versus superficial (= skin-soft tissue) revision)
Proportion of patients with aseptic revision | 1 year
  Proportion of patients with aseptic revision
Proportion of patients with implant failure | 1 year
  Proportion of patients with implant failure (any functionally affected or pain producing implant, clinically relevant abnormal laboratory test result indicating PJI, or presence of radiological signs of loosening, according to the investigator (Yes/No))
Proportion of patients with treatment failure | 1 year
  Proportion of patients with treatment failure (insufficient primary therapy or PJI relapse)
Proportion of patients with initially sufficient versus insufficient primary therapy | 1 year
  Proportion of patients with initially sufficient versus insufficient primary therapy (defined by the judgement of the investigator, based on combined clinical, laboratory, microbiological and radiological criteria, e.g. clear reduction of wound secretion)
Specific functional joint scores | 1 year
  Development and changes vs baseline of specific functional joint scores
EQ5D5L | 1 year
  EQ5D5L (in particular for 1 year follow up)
Safety and tolerability of fosfomycin (frequency of adverse events) | 1 year
  Safety and tolerability of fosfomycin will be evaluated by measuring the frequency of adverse events, including potential side effects
Pharmacokinetic profile of fosfomycin in plasma | 1 year
  Pharmacokinetic profile of fosfomycin in plasma (steady state after a single application per patient): Cmax
Pharmacokinetic profile of fosfomycin in plasma | 1 year
  Pharmacokinetic profile of fosfomycin in plasma (steady state after a single application per patient): Tmax
Pharmacokinetic profile of fosfomycin in plasma | 1 year
  Pharmacokinetic profile of fosfomycin in plasma (steady state after a single application per patient): Cmin 8 h
Pharmacokinetic profile of fosfomycin in plasma | 1 year
  Pharmacokinetic profile of fosfomycin in plasma (steady state after a single application per patient): t1/2
Pharmacokinetic profile of fosfomycin in plasma | 1 year
  Pharmacokinetic profile of fosfomycin in plasma (steady state after a single application per patient): AUC0-8
Pharmacokinetic profile of fosfomycin in plasma | 1 year
  Pharmacokinetic profile of fosfomycin in plasma (steady state after a single application per patient): extrapolated AUC0-24

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, PD Dr., Principal Investigator — Charité - Univeristätsmedizin
Locations (1):
- Charité - Univeristätsmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No